CLINICAL TRIAL: NCT04875208
Title: Latino Youth Coping With Discrimination: A Multi-Level Investigation in Micro- and Macro-Time
Brief Title: Seguimos Avanzando - Latino Youth Coping With Discrimination
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Notre Dame (Other); Fordham University (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Other Study IDs: 2020P001721
Record Dates: First submitted 2021-04-09; First posted 2021-05-06 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of this study is to investigate mediators and moderators at multiple ecological (individual, family/peer and school/neighborhood levels) and time-scale (micro- and macro-time) levels in the link between discrimination-related stressors and mental health among 340 Mexican-origin youth.

DETAILED DESCRIPTION:
The project's long-term goal is to improve the mental health of Mexican-origin youth by reducing the deleterious effects of racism, "othering," and negative neighborhood interactions. Community based collaboration will be used to recruit a sample of 340 Mexican-origin adolescents, mothers, and fathers in Indiana. The inclusion of fathers will be a valuable contribution to the literature, given the dearth of studies on Latinx fathers/stepfathers. A combination of annual surveys administered over three waves to parents and youth ("macro-time") and a 21-day daily diary ("micro-time") administered in wave 1 to youth is employed to assess important questions about how mediating and moderating processes unfold over time. Specific aims of the project include determination of within-person discrimination-related stressors that impact youth's mental health outcomes and the mechanisms of action at both micro- and macro- time levels; identification of protective factors that could help coping with discrimination related stressors and conditions under which they work; and elucidating youth, parent, and neighborhood risk factors that moderate the link between discrimination-related stressors and mental health outcomes in youth. This research is highly translational in that it will facilitate the development of more effective, culturally sensitive prevention and intervention strategies for Latinx youth and their families.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Inclusion Criteria:

* The adolescent has two eligible caregivers (as defined in the following criteria)
* The adolescent resides with at least one of the two caregivers.
* One of the caregivers is a parent or legal guardian who is eligible to give consent for the child's participation.

Caregiver Inclusion Criteria:

* Biological Parents of Mexican origin
* Legal guardians of Mexican origin
* Step-parents of Mexican origin
* A caregiver of Mexican origin identified by the parent/guardian who is 18 or older (e.g., grandparents, uncles/aunts, older siblings, godparents)

Exclusion Criteria:

* A parent reports that the adolescent has a severe learning or developmental disability which would prevent understanding/survey response

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Mexican descent adolescents between the ages of 12-15 years old (at enrollment)
  * Mexican-Origin caregivers over the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory 2nd Edition™: Self-Report Short Form [(CDI-2: SR(S)] | Time 0 (baseline)
  Youth Depression, Total score 0-24, Higher scores are worse
Children's Depression Inventory 2nd Edition™: Self-Report Short Form [(CDI-2: SR(S)] | Month 12
  Youth Depression, Total score 0-24, Higher scores are worse
Children's Depression Inventory 2nd Edition™: Self-Report Short Form [(CDI-2: SR(S)] | Month 24
  Youth Depression, Total score 0-24, Higher scores are worse
Screen for Child Anxiety Related Disorders/ [General Anxiety subscale only] (SCARED) | Time 0 (baseline)
  Youth Anxiety, Subscale Total score 0-18, Higher scores are worse
Screen for Child Anxiety Related Disorders/ [General Anxiety subscale only] (SCARED) | Month 12
  Youth Anxiety, Subscale Total score 0-18, Higher scores are worse
Screen for Child Anxiety Related Disorders/ [General Anxiety subscale only] (SCARED) | Month 24
  Youth Anxiety, Subscale Total score 0-18, Higher scores are worse
Youth Self-Report for Ages 11-18 (YSR/11-18) | Time 0 (baseline)
  Youth Psychological Symptoms
Youth Self-Report for Ages 11-18 (YSR/11-18) | Month 12
  Youth Psychological Symptoms
Youth Self-Report for Ages 11-18 (YSR/11-18) | Month 24
  Youth Psychological Symptoms
Child Behavior Checklist for Ages 6-18 (CBCL/6-18) | Time 0 (baseline)
  Adaptive Functioning
Child Behavior Checklist for Ages 6-18 (CBCL/6-18) | Month 12
  Adaptive Functioning
Child Behavior Checklist for Ages 6-18 (CBCL/6-18) | Month 24
  Adaptive Functioning
Pittsburgh Sleep Quality Index (PSQI) | Time 0 (baseline)
  Sleep Duration and Quality; Total global score (for unadapted scale) 0-21
Pittsburgh Sleep Quality Index (PSQI) | Month 12
  Sleep Duration and Quality; Total global score (for unadapted scale) 0-21
Pittsburgh Sleep Quality Index (PSQI) | Month 24
  Sleep Duration and Quality; Total global score (for unadapted scale) 0-21

CONTACTS AND LOCATIONS:
Locations (1):
- University of Notre Dame, William J. Shaw Center for Children and Families, South Bend, Indiana, United States

REFERENCES:
- [Derived] Alegria M, Cruz-Gonzalez M, Yip T, Wang L, Park IJK, Fukuda M, Valentino K, Giraldo-Santiago N, Zhen-Duan J, Alvarez K, Barrutia XA, Shrout PE. Yearly and Daily Discrimination-Related Stressors and Mexican Youth's Mental Health and Sleep: Insights From the First Wave of a Three-Wave Family Study. J Am Acad Child Adolesc Psychiatry. 2024 Nov;63(11):1134-1148. doi: 10.1016/j.jaac.2023.12.010. Epub 2024 Feb 15. PMID 38367767